CLINICAL TRIAL: NCT00938132
Title: A Clinical Trial to Evaluate the Effect of Fimarsartan on Pharmacodynamics, Pharmacokinetics, and the Safety of Warfarin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Director, Boryung Pharm Co., Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A657-BR-CT-108
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Essential Hypertension
Keywords: fimasartan; drug interaction
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Warfarin

ARMS (1):
- Fimasartan (Experimental)
  Interventions: Drug: fimasartan, warfarin

INTERVENTIONS:
Drug: fimasartan, warfarin — Warfarin(1d) Fimasartan(8d-16d) Fimasartan + Warfarin(11d)

SUMMARY:
To evaluate the effect of Fimarsartan on pharmacodynamics, pharmacokinetics, and the safety of warfarin in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 40 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan and warfarin
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism history of any serious psychological disorder
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day 3 month ago
* participation in a clinical trial during the last 2 months prior to the start of the study

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
INR AUC, INRmax, INRtmax | pre-dose, 6, 12, 24, 36, 48, 72, 96, 120, 144 h post-dose on 1 d, 11 d

SECONDARY OUTCOMES:
AUClast, AUCinf, Cmax ,Tmax, CL/F of S-warfarin and R-warfarin | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 h post-dose on 1 d, 11 d

REFERENCES:
- [Derived] Choi Y, Han H, Shin D, Lim KS, Yu KS. Comparison of the pharmacokinetics and tolerability of HCP1004 (a fixed-dose combination of naproxen and esomeprazole strontium) and VIMOVO(R) (a marketed fixed-dose combination of naproxen and esomeprazole magnesium) in healthy volunteers. Drug Des Devel Ther. 2015 Jul 31;9:4127-35. doi: 10.2147/DDDT.S86725. eCollection 2015. PMID 26257511